CLINICAL TRIAL: NCT05952843
Title: Assessment of Task Sharing Program in Family Planning and Reproductive Health in Assuit Governorate
Brief Title: Assessment of Task Sharing Program in Family Planning and Reproductive Health Services
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abo Elmakarem Alithy, Doctor, Assiut University
Other Study IDs: Task sharing
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Family Planning Services

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Support client's access to reproductive and family planning services through preferred and convenient service delivery points and overcoming barriers to accessing family planning related to the shortage of healthcare provider through strengthening the contraceptive system, capacity building of the Ministry of health personnel and training of nurses and targeting weak points in the contraceptive system through research for bridging gaps in the systems .

DETAILED DESCRIPTION:
The Sustainable Development Goals aim to meet 75% of the global demand for contraception by 2030.To meet these goals, national programs will need to bring together many components, including social and behavior change, a gender and rights perspective, commodities, and quality service provision by adequately trained health providers .

The current unmet needs for health workers that disproportionately affect low- and middle-income countries are anticipated to remain unaddressed for the next decade . It is projected that by 2030, there will be a shortage of 15 million health workers globally . In addition, inequities in the distribution of the existing health workforce within countries, with important rural versus urban differentials in both number and qualification, are worsening the coverage of services in the most deprived, yet high demand areas.

World Health Organization like many other stakeholders evolved the concept of "task sharing," as a promising strategy for addressing the critical lack of health care workers to provide reproductive, maternal, newborn care, enhancing equity in access to birth spacing methods, to obtain the desired method from their nearest service delivery point and protection against unintended pregnancies and thereby avoid costs associated with such pregnancies and of course induced / unsafe abortion.

Task sharing involves the safe expansion of tasks and procedures that are usually performed by higher-level staff to lay- and mid-level healthcare professionals such as midwives, nurses, auxiliaries, clinical officers, and community health workers, especially for the poorer segments of the society .

Task share reflects the intention to include cadres who do not normally have competencies for specific tasks to deliver them and to thereby increase levels of health care access. Moreover, it emphasizes the need for training and continued educational support of all cadres of health workers for them to undertake the tasks they are to perform .

Task shifting/sharing has been highlighted as an important strategy to optimize health worker performance in resource poor settings ; World Health Organization recommended the guidelines describe a package of technical resources for dissemination and implementation, that includes new and existing job aids, counseling tools, information sheets, sample training packages and post-training support, that must be adapted to the local context to facilitate this program .

The agencies of Family Planning Training Resource Package has been developed to be a resource for training modules on various contraceptive methods and tools. In addition, all services and guidelines should be centered in a rights-based approach that respects individual needs and preferences .

* In Burkina Faso, an increase in new users during the implementation of task sharing for family planning.
* In Ethiopia, contraceptive prevalence rate has doubled every five years from 2000 ,contraceptive prevalence rate = 6.1% to 2019 contraceptive prevalence rate = 41%. Another supporting point is the decline in total fertility rate which fell from 6.0 to 4.6 in the same period. Similarly, unmet contraceptive needs were higher in 2011 ,25.3% as compared to 2019 ,22% . From another study, anecdotal evidence health care provider observations, suggests that the back-up strategy likely positively affected client satisfaction, as they no longer needed to travel long distances to health centers to receive their method of choice.
* In Ghana, Contraception prevalence rate among married women increased from 18.6% in 2008 to 19.8% in 2014 among rural residents and from 15.1% in 2008 to 24.6% in 2014 among urban women.
* In Nigeria, Implementation of the task sharing policy for family planning increased the uptake of long-acting reversible contraception .

Egypt's population in 2022, grew by nearly 1.6 million people to reach a total of about 104.4 million at the start of this year. A baby was born every 14.4 seconds on average, according to the country's statistics agency Capmas .

The population continues to grow at a pace that presents significant challenges to social stability and the economy, especially in the governorates with the highest birth rates are mainly in Upper Egypt, including Assiut, Sohag, Qena, Minya and Beni Suef .

Egypt and United Nations Population Fund in the 10th Country Program Action Plan 2018-2022 have decided to focus on Assiut and Sohag, the 2 governorates with poor maternal health, poverty and health human resources indicators .

To stem the total fertility rate through improving the quality of voluntary family planning services and information, United States Agency for International Development works with the Egyptian government through the Ministry of Health and Population /Family Planning Sector and National Population Council . Strengthening Egypt Family Planning Program is implemented by John Snow, for technical assistance and training to decelerate Egypt's rapid population growth by reducing the unmet need of women and men for family planning counseling services and methods. Prioritizing its support in the nine governorates (Aswan, Luxor, Qena, Sohag, Assiut, Minya, Beni Suef, Fayoum, Giza ) and 11 slum areas in Cairo and Alexandria, where the need for increased access to family planning.

Accordingly, in Apri ,Strengthening Egypt's Family Planning Program , program year 2 covering the period October, 2018 to September, 2019, met the Central family planning Sector to develop a roadmap and addressing task sharing as one of Strengthening Egypt's Family Planning Program's activities related to strengthening the quality of family planning services .

That after completing the task-sharing training, nurses can provide counseling, two modern contraceptive methods to clients and others health and reproductive services , through task-share program training and about 188 nurses in 141 primary health care units in September 2022, in Egypt .

Trained nurses provide counseling and family planning services including receiving pills and injectable contraception for clients. These family planning methods contributed significantly to the country's couple year protection, this makes pills and injections the second and third most used modern contraceptive methods in Egypt among ever-married women aged 15-49 after intra uterine devices .

In Assuit governorate, the program applied in 17 health units within four districts ( Elbadarey - El qousia - Dairout - Manflout ) .

In Egypt, the public health system faces many challenges such as underfunding, low-quality care, lack of medical equipment, and shortage of qualified personnel .

Nations population Fund is partnering with reproductive health sector of the Egyptian Ministry of Health to expand family planning use to help decrease total fertility rate. The cooperation includes strengthening the contraceptive system, capacity building of the Ministry of Health personnel and training of nurses and targeting weak points in the contraceptive system through research for closing gaps in the systems .

ELIGIBILITY:
Inclusion Criteria:

* Health providers trained on program
* Maternity and family planning clinics where program has been implemented
* Women will attend maternity and family planning clinics

Exclusion Criteria:

* Not trained health providers on program
* Women not attending maternity and family planning clinics

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Trained health providers at clinics where program has been implemented.
  * Women in reproductive age who attending maternity and family planning clinics where program has been implemented and others from clinics where the program not implemented.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of implementing task sharing programs on the use and continuation of use of family planning services/ contraceptive methods. | during year 2023/2024
  revise a hard copy of rate of contraceptive use and discontinuation rate from the report of MOHP-FP sector Management Information System (MIS) will be done to compare between the achievement in the units where the program was detected and the control units.

SECONDARY OUTCOMES:
Assess the effectiveness of the program on breast examination, registration self- examination, and referral. | during year 2023/2024
  Assess the effectiveness of the program on breast examination and referral registry records will be revised
Evaluate clients' satisfaction with family planning services provided through the program. | During year 2023/2024
  Client satisfaction will be assessed using scaled questions items
Identify providers' knowledge, perception, barriers and performance in delivering task sharing program activities | during year 2023/2024
  Assessment of performance of the providers in conducting contraceptive counseling, breast examination and education sessions, safe injection and pills contraception provision, blood pressure measurement and other activities.

CONTACTS AND LOCATIONS:
Overall Officials: Faten Rabie, PHD, Study Director

REFERENCES:
- See also: Task sharing to improve access to Family Planning/Contraception.2007 — http://www.who.int
- See also: M. Guerra Arias, A. Nove, M. Michel-Schuldt, and L. de Bernis, "Current and future availability of and need for human resources for sexual, reproductive, maternal and newborn health in 41 countries in Sub-Saharan Africa," International Journal for Equi — http://www.ncbi.nlm.nih.gov
- See also: J. X. Liu, Y. Goryakin, A. Maeda, T. Bruckner, and R. Scheffler, "Global health workforce labor market projections for 2030," Human Resources for Health, vol. 15, no. 1, p. 11, 2017. — http://documents1.worldbank.org
- See also: F. Ewerling, C. G. Victora, A. Raj, C. V. N. Coll, F. Hellwig, and B. AJD, "Demand for family planning satisfied with modern methods among sexually active women in low- and middleincome countries: who is lagging behind?," Reproductive Health, vol. 15, — http://pubmed.ncbi.nlm.nih.gov
- See also: Janowitz B, Stanback J, Boyer B. Task sharing in family planning. Stud Fam Plann. 2012;43(1):57-62 — http://pubmed.ncbi.nlm.nih.gov
- See also: Millogo T, Task sharing for family planning services, Burkina Faso. Bull World Health Organ. 2019;97(11):783. — http://pubmed.ncbi.nlm.nih.gov
- See also: PMNCH/WHO, Background Paper for the Global Strategy for Women's and Children's Health: Access for All to Skilled, Motivated, and Supported Health Workers, 2010GenevaThe Partnership for Maternal, Newborn and Child Health, World Health Organization — http://platform.who.int
- See also: Kibret, M.A., Gebremedhin, L.T. Two decades of family planning in Ethiopia and the way forward to sustain hard-fought gains!. Reprod Health 19 (Suppl 1), 124 (2022). https://doi.org/10.1186/s12978-022-01435-5. — http://reproductive-health-journal.biomedcentral.com
- See also: Tilahun Y, Lew C, Belayihun B, Lulu Hagos K, Asnake M. Improving contraceptive access, use, and method mix by task sharing Implanon insertion to frontline health workers: the experience of the Integrated Family Health — http://www.ncbi.nlm.nih.gov
- See also: Independent Consultant Placide Tapsoba, Population Council, The Jagged Road to a Policy Change: Increasing Access to Family Planning using Community Health Nurses — http://uaps2015.popconf.org
- See also: Task shifting provision of contraceptive implants to community health extension workers: results of operations research in northern Nigeria. Glob Health Sci — http://dx.doi.org
- See also: Zalak, Zakarya Al, and Anne Goujon. "Exploring the fertility trend in Egypt." Demographic Research 37 (2017): 995-1030 — http://www.demographic-research.org
- See also: United Nations Population Fund 10th Country program for Egypt (2018-2022 — http://Egypt.unfpa.org
- See also: Gericke, C., Britain, K., Elmahdawy, M., & Elsisi, G. (2018, May 16). Health System in Egypt. https:///referenceworkentry/10.1007/978-1-4614-6419-8_7-1. — http://link.springer.com
- See also: United Nations Population Fund. UNFPA Egypt | Family planning. 2018 [cited 2018 Dec 18] — http://egypt.unfpa.org.